CLINICAL TRIAL: NCT05086965
Title: The Effect of Virtual Game Simulation on the Diagnosis and Goal Formation of Nursing First Year Students
Brief Title: The Effect of Virtual Game Simulation on Nursing Diagnosis and Goal Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yadigar Ordu (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor-Investigator, Yadigar Ordu, Instructor, Çankırı Karatekin University
Organization: Çankırı Karatekin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2021 - 766
Record Dates: First submitted 2021-09-29; First posted 2021-10-21 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Nursing Students
Keywords: Nursing students; Virtual game simulation; Nursing diagnosis; Nursing goal; Virtual learning; Game-based learning

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The nursing process course content prepared by the researchers in the classroom environment will be explained to the students in the control group by the researcher. After the theoretical course content is explained, the appendectomy case prepared by the researchers will be presented to the students and the case-specific nursing care plan will be explained to the students in the classroom environment by the researcher. After explaining the theoretical content and case-specific care plan preparation to the students, a test will be applied to the questions prepared according to the case sample specific to chronic obstructive pulmonary disease prepared by the researchers. Students will be asked to find the nursing diagnoses and goals specific to the presented COPD case and to prioritize the nursing diagnoses they find. Students will be graded in the order of given tests and nursing diagnoses.
- Intervention Group (Experimental): The nursing process course content prepared by the researchers will be explained to the students in the intervention group by the researcher in the classroom environment. After the theoretical course content is explained, a virtual game simulation specially developed for the appendectomy case will be played in the computer classroom of the school where the study will be conducted. At the end of the game, students will be able to see how many points they got, which questions they answered correctly and which questions they answered incorrectly. After the virtual training simulation game, students will play the virtual assessment simulation game developed for chronic obstructive pulmonary disease in the school's computer classroom. The scoring system in the game developed for COPD will be equal to the scoring system in the test that will be presented to the control group students.
  Interventions: Other: Playing the virtual game simulation

INTERVENTIONS:
Other: Playing the virtual game simulation — The virtual game simulation developed by the researchers and designed by the researchers will be played on the computer for the students of the intervention group. Virtual game simulations are virtual games developed by researchers, specific to a clinical scenario, and prepared by transferring the videos taken with an action camera to the computer environment and displaying them in two dimensions.
  Arms: Intervention Group

SUMMARY:
The study will be conducted to evaluate the effect of virtual game simulation on nursing diagnosis and goal setting skills of first year nursing students. Virtual game simulations are one of the game-based teaching methods used in nursing education with the technological developments experienced. Virtual game simulation is a two-dimensional virtual computer game based on real clinical scenarios. The use of virtual game simulations in nursing education is limited. In the researches on the subject, it is seen that the virtual game simulations of nursing students; It has been determined that it increases knowledge, psychomotor skills, motivation, satisfaction, self-efficacy, self-confidence, provides a real clinical experience, and prepares students for exams compared to a written case study. In the research, it is aimed to use virtual game simulations in nursing process teaching, which is an area where it has not been used before, and to determine its effect on the diagnosis and goal setting skills of first-year nursing students.

DETAILED DESCRIPTION:
In the study, it is aimed to evaluate the effect of virtual game simulation on the diagnosis and goal setting skills of first year nursing students. For this purpose, the research will be conducted with first-year nursing students who meet the criteria for participation in the research and agree to participate in the study. Ethics committee permission and institutional permission were obtained from the relevant institution before starting the study. In the study, students will be randomly divided into control and intervention groups. Randomization and evaluation of the results will be performed by those other than the researchers, thus providing triple blinding in the study. First of all, the theoretical course content of the nursing process prepared by the researchers in the classroom environment will be explained to the control group students and the intervention group students. Then, it will be applied to the control group students with pencil and paper in the Chronic obstructive pulmonary disease case, which consists of an educational appendectomy document and an evaluation test in the classroom environment. The students of the intervention group will play the virtual game simulation in the computer classroom of the school where the study will be conducted, in the same way as the cases applied to the control group. The effect of the simulation game on diagnosis and goal creation will be determined. At the end of the study, simulation games will be played to the students in the control group and all other students in the class who were not included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Taking the Nursing Fundamentals II course,
* All students who accept to participate in the study will be accepted.

Exclusion Criteria:

* Retaking the Nursing Fundamentals II course,
* Graduated from Health Vocational High School,
* Having any previous experience in the nursing process,
* Having difficulty in understanding and speaking Turkish,
* Coming with horizontal and vertical transition,
* Students who do not volunteer to participate in the research will not be included in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-24 (Actual)

PRIMARY OUTCOMES:
Knowledge of determining the correct case-specific nursing diagnosis | 1 month
  The percentage of students in the experimental and control groups who determined the correct nursing diagnosis
Knowledge of determining the correct case-specific patient target | 1 month
  The percentages of students in the experimental and control groups determining the correct patient goals

CONTACTS AND LOCATIONS:
Locations (1):
- Cankiri, Çankırı, Turkey (Türkiye)